CLINICAL TRIAL: NCT01989754
Title: A Randomized, Multicenter, Double-Blind, Parallel, Placebo-Controlled Study of the Effects of Canagliflozin on Renal Endpoints in Adult Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study of the Effects of Canagliflozin (JNJ-28431754) on Renal Endpoints in Adult Participants With Type 2 Diabetes Mellitus
Acronym: CANVAS-R
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: The George Institute for Global Health, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR102647; 2013-003050-25 (EudraCT Number); 28431754DIA4003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-10-17; First posted 2013-11-21 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2; Albuminuria
Keywords: Albuminuria; Canagliflozin; Cardiovascular outcomes; Type 2 Diabetes Mellitus; T2DM; JNJ-28431754; Antihyperglycemic Agent
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Albuminuria | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (2):
- Canagliflozin (JNJ-28431754) (Experimental): Each patient will receive canagliflozin (JNJ-28431754) 100 mg once daily during the first 13 weeks, then the dose may be increased to 300 mg once daily.
  Interventions: Drug: Canagliflozin, 100 mg; Drug: Canagliflozin, 300 mg
- Placebo (Placebo Comparator): Each patient will receive placebo (inactive medication) once daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — One placebo capsule taken orally (by mouth) once daily for 156 weeks
  Arms: Placebo
Drug: Canagliflozin, 100 mg — One 100 mg capsule taken orally (by mouth) once daily
  Arms: Canagliflozin (JNJ-28431754)
Drug: Canagliflozin, 300 mg — One 300 mg capsule taken orally (by mouth) once daily
  Arms: Canagliflozin (JNJ-28431754)

SUMMARY:
The purpose of this study is to assess the effect of canagliflozin compared to placebo on progression of albuminuria in participants with Type 2 Diabetes Mellitus receiving standard care but with inadequate glycemic control and at elevated risk of cardiovascular events.

DETAILED DESCRIPTION:
The study will be conducted in adult participants with Type 2 Diabetes Mellitus (T2DM), receiving standard of care for hyperglycemia and cardiovascular (CV) risk factors, who have either a history of a prior CV event or 2 or more risk factors for a CV event. Participants will be randomly assigned in a 1:1 ratio to canagliflozin or matching placebo to be taken once daily. Canagliflozin will be provided at a dose of 100 mg/day through Week 13 and then increased at the discretion of the investigator to a dose of 300 mg/day, if the participant requires additional glycemic control and is tolerating the 100 mg dose.

The study consists of a 2-week screening period and a double-blind treatment period lasting between 78 and 156 weeks; study completion is targeted for when the last subject randomized has approximately 78 weeks of follow-up or when 688 major adverse cardiovascular events are accumulated between CANVAS and CANVAS-R. A total of 5,700 participants are targeted to be recruited into the study. Participants can be either drug naïve to antihyperglycemic agents, using monotherapy, or using combination of antihyperglycemic therapy for the control of blood glucose levels.

The completion target was reached in February 2017.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of type 2 diabetes mellitus
* Must have inadequate diabetes control (as defined by glycosylated hemoglobin level >=7.0% to <=10.5% at screening)
* Greater than or equal to (>=) 30 yrs old with history of cardiovascular (CV) event, or >= 50 yrs old with high risk of CV events
* Must be either not on antihyperglycemic agents (AHA) therapy, or on AHA monotherapy, or combination AHA therapy with any approved agent for the control of blood glucose levels.

Exclusion Criteria

* History of diabetic ketoacidosis, type 1 diabetes mellitus, pancreas or beta-cell transplantation, or diabetes secondary to pancreatitis or pancreatectomy
* History of one or more severe hypoglycemic episode within 6 months before screening
* History of hereditary glucose-galactose malabsorption or primary renal glucosuria
* Ongoing, inadequately controlled thyroid disorder
* Renal disease that required treatment with immunosuppressive therapy or a history of chronic dialysis or renal transplant
* Myocardial infarction, unstable angina, revascularization procedure, or cerebrovascular accident within 3 months before screening.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5813 (Actual)
Dates: Start 2014-01-16 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (342):
- United States (57):
  - Little Rock, Arkansas
  - Carmichael, California
  - Concord, California
  - Pismo Beach, California
  - Roseville, California
  - Thousand Oaks, California
  - Denver, Colorado
  - Hollywood, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Opa-locka, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Tampa, Florida
  - Meridian, Idaho
  - Chicago, Illinois
  - Valparaiso, Indiana
  - Topeka, Kansas
  - Louisville, Kentucky
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Elkridge, Maryland
  - Flint, Michigan
  - Picayune, Mississippi
  - Kansas City, Missouri
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Cornelius, North Carolina
  - Hickory, North Carolina
  - Mooresville, North Carolina
  - Canal Fulton, Ohio
  - Franklin, Ohio
  - Mason, Ohio
  - Oklahoma City, Oklahoma
  - Beaver, Pennsylvania
  - Levittown, Pennsylvania
  - Norristown, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Tipton, Pennsylvania
  - Greer, South Carolina
  - Jefferson City, Tennessee
  - Austin, Texas
  - Pearland, Texas
  - Bountiful, Utah
  - Draper, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - South Burlington, Vermont
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Virginia Beach, Virginia
  - Spokane, Washington
  - Milwaukee, Wisconsin
  - Wauwatosa, Wisconsin
- Argentina (7):
  - Buenos Aires
  - Ciudad de Buenos Aires
  - Córdoba
  - Mar del Plata
  - Morón
  - Rosario
  - Zarate, Buenos Aires
- Australia (12):
  - Box Hill
  - Cairns
  - Daw Park
  - Freemantle
  - Liverpool
  - Melbourne
  - Newcastle
  - Sherwood
  - Sydney
  - Tasmania
  - Woden
  - Woolloongabba
- Belgium (12):
  - Bonheiden
  - Bruges
  - Edegem
  - Ghent
  - La Louvière
  - Leuven
  - Liège
  - Liÿge
  - Merksem
  - Ransart
  - Roeselare
  - Tessenderlo
- Brazil (12):
  - Belém
  - Belo Horizonte
  - Campinas
  - Caxias do Sul
  - Curitiba
  - Fortaleza
  - Mogi das Cruzes
  - Passo Fundo
  - Porto Alegre
  - Rio de Janeiro
  - São José do Rio Preto
  - São Paulo
- Canada (16):
  - Coquitlam, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - Guelph, Ontario
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Sarnia, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
  - Laval, Quebec
  - Lévis, Quebec
  - Québec, Quebec
  - Saint Marc Des Carriéres, Quebec
  - Sherbrooke, Quebec
  - Westmont, Quebec
  - Saskatoon, Saskatchewan
- China (6):
  - Baotou
  - Beijing
  - Hangzhou
  - Jinan
  - Shenyang
  - Wuxi
- Czechia (5):
  - Beroun
  - Ostrava
  - Pilsen
  - Prague
  - Znojmo
- France (10):
  - Amiens
  - Bois-Guillaume
  - Bordeaux
  - Dijon
  - Grenoble
  - La Rochelle
  - Le Creusot
  - Narbonne
  - Paris
  - Poitiers
- Germany (12):
  - Aschaffenburg
  - Aßlar
  - Bad Oeynhausen
  - Dortmund
  - Dresden
  - Freiburg im Breisgau
  - Hanover
  - Kassel
  - Mainz
  - Neuwied
  - Saarbrücken
  - Villingen-Schwenningen
- Hungary (11):
  - Balatonfüred
  - Budapest
  - Dunaújváros
  - Eger
  - Kecskemét
  - Nagykanizsa
  - Pécs
  - Székesfehérvár
  - Szikszó
  - Szombathely
  - Zalaegerszeg
- Italy (13):
  - *Osenza*
  - Arenzano
  - Bologna
  - Catanzaro
  - Chieri (Torino)
  - Florence
  - Messina
  - Milan
  - Napoli
  - Ravenna
  - Roma
  - Sesto San Giovanni (Milano)
  - Verona
- Malaysia (7):
  - Batu Caves
  - George Town
  - Ipoh
  - Kelantan
  - Kota Bharu
  - Kuala Lumpur
  - Kuching
- Mexico (10):
  - Aguascalientes
  - Celaya
  - Cuernavaca
  - Culiacán
  - Guadalajara
  - México
  - Pachuca
  - Querétaro
  - San Luis Potosí City
  - Tampico
- Netherlands (21):
  - Almelo
  - Almere Stad
  - Amersfoort
  - Amsterdam
  - Dordrecht
  - Eindhoven
  - Groningen
  - Hardenberg
  - Hoogeveen
  - Hoogezand
  - Kloosterhaar
  - Leiden
  - Meppel
  - Poortvliet
  - Rotterdam
  - Utrecht
  - Velp
  - Waalwijk
  - Wamel
  - Zoetermeer
  - Zwijndrecht
- New Zealand (7):
  - Auckland
  - Christchurch
  - Newtown
  - Palmerston North
  - Rotorua
  - Tauranga
  - Wellington
- Poland (13):
  - Bialystok
  - Bydgoszcz
  - Chrzanów
  - Gdansk
  - Grodzisk Mazowiecki
  - Katowice
  - Krakow
  - Lublin
  - Oświęcim
  - Torun
  - Tychy
  - Warsaw
  - Wroclaw
- Puerto Rico (2):
  - Ponce Pr
  - Trujillo Alto
- Russia (15):
  - Arkhangelsk
  - Barnaul
  - Chelyabinsk
  - Kemerovo
  - Nizhny Novgorod
  - Penza
  - Rostov-on-Don
  - Saint Petersburg
  - Samara
  - Saratov
  - Smolensk
  - Syktyvkar
  - Tyumen
  - Vsevolzhsk
  - Yaroslavl
- South Korea (15):
  - Ansan
  - Bucheon-si
  - Busan
  - Changwon
  - Cheongju-si
  - Daegu
  - Gyeonggi-do
  - Iksan
  - Incheon
  - Jeonju
  - Seongnam-si
  - Seoul
  - Suwon
  - Ulsan
  - Wŏnju
- Spain (24):
  - A Coruña
  - Alcalá de Henares
  - Alicante
  - Almería
  - Alzira
  - Barcelona
  - Ciudad Real
  - Córdoba
  - Ferrol
  - Figueres
  - Galdakao
  - Madrid
  - Málaga
  - Móstoles
  - Palma de Mallorca
  - Sabadell
  - San Sebastián de los Reyes
  - Sant Joan d'Alacant
  - Santa Cruz de Tenerife
  - Santiago de Compostela
  - Segovia
  - Seville
  - Valencia
  - Viladecans
- Sweden (12):
  - Borås
  - Gothenburg
  - Helsingborg
  - Karlstad
  - Linköping
  - Lund
  - Malmo
  - Stockholm
  - Uddevalla
  - Uppsala
  - Vällingby
  - Västra Frölunda
- Taiwan (6):
  - Kaohsiung County
  - Taichung
  - Tainan
  - Taipei
  - Tiachung
  - Xindian
- Ukraine (18):
  - Cherkasy
  - Chernivtsy
  - Dnipropetrovsk
  - Ivan-Frankivsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Lviv
  - Odesa
  - Poltava
  - Sumy
  - Ternopil
  - Uzhhorod
  - Vinnitsa
  - Vinnytsia
  - Zaporizhzhia
  - Zaporizhzhya
- United Kingdom (19):
  - Addlestone
  - Belfast
  - Birmingham
  - Blackburn
  - Bristol
  - Bury St Edmunds
  - Chesterfield
  - Derby
  - Doncaster
  - Ipswich
  - Leicester
  - Liverpool
  - Manchester
  - Salford
  - Taunton
  - Torquay
  - Truro
  - Wellingborough
  - Welwyn Garden City

REFERENCES:
- [Derived] Januzzi JLJ, Sattar N, Vaduganathan M, Magaret CA, Rhyne RF, Liu Y, Masson S, Butler J, Hansen MK. A validated multivariable machine learning model to predict cardio-kidney risk in diabetic kidney disease. Cardiovasc Diabetol. 2025 May 15;24(1):213. doi: 10.1186/s12933-025-02779-5. PMID 40375260
- [Derived] Doi Y, Hamano T, Yamaguchi O, Isaka Y. Canagliflozin may increase thromboembolic events in males with erythrocytosis but not in females. Blood Adv. 2025 Jul 8;9(13):3202-3212. doi: 10.1182/bloodadvances.2025016320. PMID 40239057
- [Derived] Nguyen TN, Yu J, Perkovic V, Jardine M, Mahaffey KW, Chow CK, Arnott C, Lindley RI. The Efficacy and Safety of Canagliflozin by Frailty Status in Participants of the CANVAS and CREDENCE Trials. J Am Geriatr Soc. 2025 Jun;73(6):1787-1796. doi: 10.1111/jgs.19444. Epub 2025 Mar 19. PMID 40105285
- [Derived] Vaduganathan M, Cannon CP, Jardine MJ, Heerspink HJL, Arnott C, Neuen BL, Sarraju A, Gogate J, Seufert J, Neal B, Perkovic V, Mahaffey KW, Kosiborod MN. Effects of canagliflozin on total heart failure events across the kidney function spectrum: Participant-level pooled analysis from the CANVAS Program and CREDENCE trial. Eur J Heart Fail. 2024 Sep;26(9):1967-1975. doi: 10.1002/ejhf.3292. Epub 2024 Jun 26. PMID 38932575
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Sharma A, Razaghizad A, Joury A, Levin A, Bajaj HS, Mancini GBJ, Wong NC, Slee A, Ang FG, Rapattoni W, Neuen BL, Arnott C, Perkovic V, Mahaffey KW. Primary and Secondary Cardiovascular and Kidney Prevention With Canagliflozin: Insights From the CANVAS Program and CREDENCE Trial. J Am Heart Assoc. 2024 Feb 6;13(3):e031586. doi: 10.1161/JAHA.123.031586. Epub 2024 Jan 19. PMID 38240199
- [Derived] Yu J, Sweeting AN, Gianacas C, Houston L, Lee V, Fletcher RA, Perkovic V, Li Q, Neuen BL, Berwanger O, Heerspink HJL, de Zeeuw D, Arnott C. The effects of canagliflozin in type 2 diabetes in subgroups defined by population-specific body mass index: Insights from the CANVAS Program and CREDENCE trial. Diabetes Obes Metab. 2023 Dec;25(12):3724-3735. doi: 10.1111/dom.15267. Epub 2023 Sep 6. PMID 37671609
- [Derived] Fletcher RA, Arnott C, Rockenschaub P, Schutte AE, Carpenter L, Vaduganathan M, Agarwal R, Bakris G, Chang TI, Heerspink HJL, Jardine MJ, Mahaffey KW, Neal B, Pollock C, Jun M, Rodgers A, Perkovic V, Neuen BL. Canagliflozin, Blood Pressure Variability, and Risk of Cardiovascular, Kidney, and Mortality Outcomes: Pooled Individual Participant Data From the CANVAS and CREDENCE Trials. J Am Heart Assoc. 2023 Jul 4;12(13):e028516. doi: 10.1161/JAHA.122.028516. Epub 2023 Jun 22. PMID 37345834
- [Derived] Borisov AN, Kutz A, Christ ER, Heim MH, Ebrahimi F. Canagliflozin and Metabolic Associated Fatty Liver Disease in Patients With Diabetes Mellitus: New Insights From CANVAS. J Clin Endocrinol Metab. 2023 Oct 18;108(11):2940-2949. doi: 10.1210/clinem/dgad249. PMID 37149821
- [Derived] Ferrannini G, Pollock C, Natali A, Yavin Y, Mahaffey KW, Ferrannini E. Extremes of both weight gain and weight loss are associated with increased incidence of heart failure and cardiovascular death: evidence from the CANVAS Program and CREDENCE. Cardiovasc Diabetol. 2023 Apr 29;22(1):100. doi: 10.1186/s12933-023-01832-5. PMID 37120538
- [Derived] Nunes JC, Yu J, Arnott C, Jardine MJ, Perkovic V, Mahaffey KW. Canagliflozin, mental health adverse events and diabetes: Exploratory analysis of the CREDENCE trial and CANVAS Program. Diabetes Obes Metab. 2022 Dec;24(12):2459-2464. doi: 10.1111/dom.14832. Epub 2022 Aug 19. No abstract available. PMID 35938182
- [Derived] Young TK, Li JW, Kang A, Heerspink HJL, Hockham C, Arnott C, Neuen BL, Zoungas S, Mahaffey KW, Perkovic V, de Zeeuw D, Fulcher G, Neal B, Jardine M. Effects of canagliflozin compared with placebo on major adverse cardiovascular and kidney events in patient groups with different baseline levels of HbA1c, disease duration and treatment intensity: results from the CANVAS Program. Diabetologia. 2021 Nov;64(11):2402-2414. doi: 10.1007/s00125-021-05524-1. Epub 2021 Aug 26. PMID 34448033
- [Derived] Yu J, Li J, Leaver PJ, Arnott C, Huffman MD, Udell JA, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Rosenthal N, Neal B, Figtree GA. Effects of canagliflozin on myocardial infarction: a post hoc analysis of the CANVAS programme and CREDENCE trial. Cardiovasc Res. 2022 Mar 16;118(4):1103-1114. doi: 10.1093/cvr/cvab128. PMID 33826709
- [Derived] Yu J, Arnott C, Neuen BL, Heersprink HL, Mahaffey KW, Cannon CP, Khan SS, Baldridge AS, Shah SJ, Huang Y, Li C, Figtree GA, Perkovic V, Jardine MJ, Neal B, Huffman MD. Cardiovascular and renal outcomes with canagliflozin according to baseline diuretic use: a post hoc analysis from the CANVAS Program. ESC Heart Fail. 2021 Apr;8(2):1482-1493. doi: 10.1002/ehf2.13236. Epub 2021 Feb 17. PMID 33595905
- [Derived] Neuen BL, Ohkuma T, Neal B, Matthews DR, de Zeeuw D, Mahaffey KW, Fulcher G, Blais J, Li Q, Jardine MJ, Perkovic V, Wheeler DC. Relative and Absolute Risk Reductions in Cardiovascular and Kidney Outcomes With Canagliflozin Across KDIGO Risk Categories: Findings From the CANVAS Program. Am J Kidney Dis. 2021 Jan;77(1):23-34.e1. doi: 10.1053/j.ajkd.2020.06.018. Epub 2020 Sep 21. PMID 32971190
- [Derived] Oshima M, Neal B, Toyama T, Ohkuma T, Li Q, de Zeeuw D, Heerspink HJL, Mahaffey KW, Fulcher G, Canovatchel W, Matthews DR, Perkovic V. Different eGFR Decline Thresholds and Renal Effects of Canagliflozin: Data from the CANVAS Program. J Am Soc Nephrol. 2020 Oct;31(10):2446-2456. doi: 10.1681/ASN.2019121312. Epub 2020 Jul 21. PMID 32694216
- [Derived] Matthews DR, Wysham C, Davies M, Slee A, Alba M, Lee M, Perkovic V, Mahaffey KW, Neal B. Effects of canagliflozin on initiation of insulin and other antihyperglycaemic agents in the CANVAS Program. Diabetes Obes Metab. 2020 Nov;22(11):2199-2203. doi: 10.1111/dom.14143. Epub 2020 Aug 24. PMID 32691499
- [Derived] Li J, Woodward M, Perkovic V, Figtree GA, Heerspink HJL, Mahaffey KW, de Zeeuw D, Vercruysse F, Shaw W, Matthews DR, Neal B. Mediators of the Effects of Canagliflozin on Heart Failure in Patients With Type 2 Diabetes. JACC Heart Fail. 2020 Jan;8(1):57-66. doi: 10.1016/j.jchf.2019.08.004. Epub 2019 Oct 29. PMID 31676303
- [Derived] Zhou Z, Jardine M, Perkovic V, Matthews DR, Mahaffey KW, de Zeeuw D, Fulcher G, Desai M, Oh R, Simpson R, Watts NB, Neal B. Canagliflozin and fracture risk in individuals with type 2 diabetes: results from the CANVAS Program. Diabetologia. 2019 Oct;62(10):1854-1867. doi: 10.1007/s00125-019-4955-5. Epub 2019 Aug 10. PMID 31399845
- [Derived] Figtree GA, Radholm K, Barrett TD, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Matthews DR, Shaw W, Neal B. Effects of Canagliflozin on Heart Failure Outcomes Associated With Preserved and Reduced Ejection Fraction in Type 2 Diabetes Mellitus. Circulation. 2019 May 28;139(22):2591-2593. doi: 10.1161/CIRCULATIONAHA.119.040057. Epub 2019 Mar 17. No abstract available. PMID 30882240
- [Derived] Zhou Z, Lindley RI, Radholm K, Jenkins B, Watson J, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Shaw W, Oh R, Desai M, Matthews DR, Neal B. Canagliflozin and Stroke in Type 2 Diabetes Mellitus. Stroke. 2019 Feb;50(2):396-404. doi: 10.1161/STROKEAHA.118.023009. PMID 30591006
- [Derived] Neuen BL, Ohkuma T, Neal B, Matthews DR, de Zeeuw D, Mahaffey KW, Fulcher G, Desai M, Li Q, Deng H, Rosenthal N, Jardine MJ, Bakris G, Perkovic V. Cardiovascular and Renal Outcomes With Canagliflozin According to Baseline Kidney Function. Circulation. 2018 Oct 9;138(15):1537-1550. doi: 10.1161/CIRCULATIONAHA.118.035901. PMID 29941478
- [Derived] Perkovic V, de Zeeuw D, Mahaffey KW, Fulcher G, Erondu N, Shaw W, Barrett TD, Weidner-Wells M, Deng H, Matthews DR, Neal B. Canagliflozin and renal outcomes in type 2 diabetes: results from the CANVAS Program randomised clinical trials. Lancet Diabetes Endocrinol. 2018 Sep;6(9):691-704. doi: 10.1016/S2213-8587(18)30141-4. Epub 2018 Jun 21. PMID 29937267
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Eligibility varies among the 4 sodium-glucose cotransporter-2 inhibitor cardiovascular outcomes trials: implications for the general type 2 diabetes US population. Am J Manag Care. 2018 Apr;24(8 Suppl):S138-S145. PMID 29693360
- [Derived] Radholm K, Figtree G, Perkovic V, Solomon SD, Mahaffey KW, de Zeeuw D, Fulcher G, Barrett TD, Shaw W, Desai M, Matthews DR, Neal B. Canagliflozin and Heart Failure in Type 2 Diabetes Mellitus: Results From the CANVAS Program. Circulation. 2018 Jul 31;138(5):458-468. doi: 10.1161/CIRCULATIONAHA.118.034222. PMID 29526832
- [Derived] Mahaffey KW, Neal B, Perkovic V, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Fabbrini E, Sun T, Li Q, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin for Primary and Secondary Prevention of Cardiovascular Events: Results From the CANVAS Program (Canagliflozin Cardiovascular Assessment Study). Circulation. 2018 Jan 23;137(4):323-334. doi: 10.1161/CIRCULATIONAHA.117.032038. Epub 2017 Nov 13. PMID 29133604
- [Derived] Neal B, Perkovic V, Mahaffey KW, de Zeeuw D, Fulcher G, Erondu N, Shaw W, Law G, Desai M, Matthews DR; CANVAS Program Collaborative Group. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017 Aug 17;377(7):644-657. doi: 10.1056/NEJMoa1611925. Epub 2017 Jun 12. PMID 28605608

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 5,813 participants were randomized. However, 1 participant was randomized twice and only the first randomization was included in the Intent-to-treat (ITT) analysis set. Thus 2,905 and 2,907 participants were randomly assigned to the placebo and canagliflozin groups in the ITT analysis set, respectively.
Groups:
- Placebo (Placebo): Participants received one capsule of matching placebo orally once daily for the duration of the study or until early discontinuation from treatment.
- Canagliflozin (Experimental): Participants received canagliflozin (JNJ-28431754) 100 milligram (mg) once daily during the first 13 weeks, then the dose was increased to 300 mg once daily (if the participant required additional glycemic control, provided the 100-mg dose was well tolerated).
Period: Overall Study
Arm/Group | Placebo (Placebo) | Canagliflozin (Experimental)
Started | 2905 | 2907
Treated | 2903 | 2904
Completed | 2866 (Participants who died are included in this category.) | 2872 (Participants who died are included in this category.)
Not Completed | 39 | 35
Not completed — Withdrawal by Subject | 10 | 14
Not completed — Lost to Follow-up | 28 | 20
Not completed — Closed Site | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Placebo) | Canagliflozin (Experimental) | Total
Number analyzed (Participants) | 2905 | 2907 | 5812
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.28) | 63.9 (8.42) | 64 (8.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1111 | 1053 | 2164
  Male | 1794 | 1854 | 3648
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 586 | 604 | 1190
  Not Hispanic or Latino | 2303 | 2290 | 4593
  Unknown or Not Reported | 16 | 13 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 14 | 33
  Asian | 245 | 244 | 489
  Native Hawaiian or Other Pacific Islander | 09 | 08 | 17
  Black or African American | 125 | 106 | 231
  White | 2372 | 2393 | 4765
  More than one race | 10 | 09 | 19
  Unknown or Not Reported | 125 | 133 | 258
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 245 | 244 | 489
  Black or African American | 125 | 106 | 231
  Hispanic or Latino | 407 | 437 | 844
  Other | 174 | 172 | 346
  White Non-Hispanic | 1954 | 1948 | 3902
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 146 | 159 | 305
  AUSTRALIA | 58 | 51 | 109
  BELGIUM | 86 | 66 | 152
  BRAZIL | 277 | 272 | 549
  CANADA | 136 | 146 | 282
  CHINA | 46 | 46 | 92
  CZECH REPUBLIC | 67 | 72 | 139
  FRANCE | 69 | 55 | 124
  GERMANY | 46 | 55 | 101
  HUNGARY | 82 | 97 | 179
  ITALY | 49 | 49 | 98
  MALAYSIA | 50 | 42 | 92
  MEXICO | 118 | 110 | 228
  NETHERLANDS | 117 | 132 | 249
  NEW ZEALAND | 49 | 56 | 105
  POLAND | 186 | 177 | 363
  RUSSIAN FEDERATION | 213 | 199 | 412
  SOUTH KOREA | 73 | 94 | 167
  SPAIN | 247 | 249 | 496
  SWEDEN | 118 | 103 | 221
  TAIWAN | 44 | 32 | 76
  UKRAINE | 213 | 236 | 449
  UNITED KINGDOM | 78 | 73 | 151
  UNITED STATES | 337 | 336 | 673

OUTCOME MEASURES:

1. Primary Outcome: Progression of Albuminuria
Description: Progression defined as the development of micro-albuminuria (Urine Albumin Creatinine Ratio [UACR] 30 to 300 milligram per gram [mg/g]) or macroalbuminuria (Albumin/creatinine ratio [ACR] of greater than [>] 300 mg/g) in a participant with baseline normoalbuminuria (ACR less than [<] 30 mg/g) or the development of macro-albuminuria in a participant with baseline microalbuminuria with an ACR increase greater than or equal to (>=) 30 percent from baseline. Participants with macroalbuminuria at baseline (ACR>300 mg/g) were excluded from the analysis. Event rate was estimated based on the time to the first occurrence of the event.
Time Frame: Up to 3 years
Population: The intent to treat (ITT) population included all participants who were randomized. Here 'N' signifies number of participants who were evaluable for this endpoint.
Measure: Number; unit: Events per 1000 patient-year
Groups:
- Placebo: Participants received one capsule of matching placebo orally once daily for the duration of the study or until early discontinuation from treatment.
Arm/Group | Placebo | Canagliflozin (Experimental)
Number analyzed (Participants) | 2905 | 2907
Events per 1000 patient-year | 153.01 | 99.80
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin (Experimental); Test type: Superiority; p < .0001, Cox proportional hazard method; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.57 to 0.73]

2. Secondary Outcome: Composite of Cardiovascular (CV) Death Events or Hospitalization for Heart Failure
Description: Analyses were using adjudicated events, that is (i.e.) CV death events or hospitalization due to heart failure, and adjudication of these outcomes by the Endpoint Adjudication Committee (EAC) were done in a blinded fashion. Event rate was estimated based on the time to the first occurrence of the event.
Time Frame: Approximately 3 years
Population: ITT population included all participants who were randomized.
Measure: Number; unit: Events per 1000 patient-years
Arm/Group | Placebo | Canagliflozin (Experimental)
Number analyzed (Participants) | 2905 | 2907
Events per 1000 patient-years | 21.91 | 15.85
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin (Experimental); Test type: Superiority; p = 0.0148, Stratified Cox proportional hazard; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.55 to 0.94]

3. Secondary Outcome: Cardiovascular (CV) Death
Description: Analyses were using adjudicated events, i.e. CV death events, and adjudication of these outcomes by the Endpoint Adjudication Committee (EAC) were done in a blinded fashion. Event rate was estimated based on the time to the first occurrence of the event.
Time Frame: Approximately 3 years
Population: ITT population included all participants who were randomized.
Measure: Number; unit: Events per 1000 patient-years
Arm/Group | Placebo | Canagliflozin (Experimental)
Number analyzed (Participants) | 2905 | 2907
Events per 1000 patient-years | 11.60 | 10.06
Statistical Analysis 1: Comparison: Placebo vs Canagliflozin (Experimental); Test type: Superiority; p = 0.4067, Stratified Cox proportional hazard; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.61 to 1.22]

ADVERSE EVENTS:
Time Frame: Approximately 3 years
Description: On-treatment analysis set included all randomized participants who were treated and received at least 1 dose of study drug. The number of deaths (all causes) reported here is adjudicated death that occurred within 30 days of the last dose of the study drug.
Arm/Group | Placebo (Placebo) | Canagliflozin (Experimental)
All-Cause Mortality (participants affected / at risk) | 71/2903 | 68/2904
Serious Adverse Events (participants affected / at risk) | 775/2903 | 714/2904
Other Adverse Events (participants affected / at risk) | 25/2903 | 94/2904
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo) (N=2903) | Canagliflozin (Experimental) (N=2904)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2 | 1
Polycythaemia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute Coronary Syndrome (Cardiac disorders) | 11 | 4
Acute Left Ventricular Failure (Cardiac disorders) | 1 | 1
Acute Myocardial Infarction (Cardiac disorders) | 26 | 32
Adams-Stokes Syndrome (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 33 | 22
Angina Unstable (Cardiac disorders) | 42 | 42
Aortic Valve Disease (Cardiac disorders) | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 2
Arteriosclerosis Coronary Artery (Cardiac disorders) | 5 | 3
Atrial Fibrillation (Cardiac disorders) | 18 | 14
Atrial Flutter (Cardiac disorders) | 7 | 5
Atrial Tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 1 | 3
Atrioventricular Block Second Degree (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 2
Cardiac Arrest (Cardiac disorders) | 9 | 5
Cardiac Disorder (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 41 | 19
Cardiac Failure Acute (Cardiac disorders) | 3 | 2
Cardiac Failure Chronic (Cardiac disorders) | 3 | 4
Cardiac Failure Congestive (Cardiac disorders) | 18 | 11
Cardiac Valve Disease (Cardiac disorders) | 2 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 1
Cardiogenic Shock (Cardiac disorders) | 2 | 0
Cardiopulmonary Failure (Cardiac disorders) | 0 | 1
Conduction Disorder (Cardiac disorders) | 2 | 0
Congestive Cardiomyopathy (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 29 | 34
Coronary Artery Insufficiency (Cardiac disorders) | 0 | 1
Coronary Artery Occlusion (Cardiac disorders) | 3 | 4
Coronary Artery Stenosis (Cardiac disorders) | 8 | 5
Diabetic Cardiomyopathy (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 4 | 1
Left Ventricular Dysfunction (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 1
Mitral Valve Stenosis (Cardiac disorders) | 0 | 1
Myocardial Fibrosis (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 24 | 31
Myocardial Ischaemia (Cardiac disorders) | 9 | 7
Pericardial Effusion (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 3 | 0
Prinzmetal Angina (Cardiac disorders) | 1 | 0
Right Ventricular Failure (Cardiac disorders) | 2 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 4 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Tricuspid Valve Incompetence (Cardiac disorders) | 0 | 1
Ventricular Arrhythmia (Cardiac disorders) | 1 | 0
Ventricular Asystole (Cardiac disorders) | 1 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 1
Ventricular Fibrillation (Cardiac disorders) | 0 | 2
Ventricular Tachycardia (Cardiac disorders) | 2 | 1
Haematotympanum (Ear and labyrinth disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1
Basedow's Disease (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 2 | 0
Hyperparathyroidism Primary (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 1 | 0
Amaurosis Fugax (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 10
Diabetic Retinopathy (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 2
Eye Haemorrhage (Eye disorders) | 1 | 0
Eye Pain (Eye disorders) | 1 | 0
Eyelid Ptosis (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Macular Fibrosis (Eye disorders) | 0 | 1
Retinal Artery Occlusion (Eye disorders) | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 1 | 0
Abdominal Hernia (Gastrointestinal disorders) | 3 | 0
Abdominal Pain (Gastrointestinal disorders) | 5 | 2
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Anal Fistula (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Barrett's Oesophagus (Gastrointestinal disorders) | 1 | 0
Bowel Movement Irregularity (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 1
Colitis Microscopic (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Colonic Pseudo-Obstruction (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Diverticular Perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 2
Diverticulum Intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 | 0
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Polyps (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 3
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Impaired Gastric Emptying (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 4 | 2
Intestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 3 | 0
Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Large Intestine Perforation (Gastrointestinal disorders) | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1
Melaena (Gastrointestinal disorders) | 0 | 2
Mesenteric Arterial Occlusion (Gastrointestinal disorders) | 0 | 1
Mesenteric Vein Thrombosis (Gastrointestinal disorders) | 2 | 0
Oesophageal Obstruction (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 2 | 3
Peptic Ulcer (Gastrointestinal disorders) | 1 | 2
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Rectal Tenesmus (Gastrointestinal disorders) | 1 | 0
Salivary Gland Calculus (Gastrointestinal disorders) | 0 | 1
Salivary Gland Fistula (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 2
Swollen Tongue (Gastrointestinal disorders) | 1 | 0
Tooth Disorder (Gastrointestinal disorders) | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 1 | 6
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 3
Volvulus (Gastrointestinal disorders) | 1 | 0
Adverse Drug Reaction (General disorders) | 1 | 1
Cardiac Death (General disorders) | 1 | 0
Chest Discomfort (General disorders) | 2 | 0
Chest Pain (General disorders) | 17 | 22
Complication Associated with Device (General disorders) | 0 | 1
Cyst (General disorders) | 1 | 0
Death (General disorders) | 7 | 5
Drug Intolerance (General disorders) | 0 | 1
Gait Disturbance (General disorders) | 0 | 1
Generalised Oedema (General disorders) | 1 | 0
Impaired Healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 1
Non-Cardiac Chest Pain (General disorders) | 7 | 9
Oedema Peripheral (General disorders) | 2 | 0
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Sudden Cardiac Death (General disorders) | 1 | 0
Sudden Death (General disorders) | 6 | 6
Vascular Stent Restenosis (General disorders) | 0 | 1
Vascular Stent Thrombosis (General disorders) | 1 | 0
Bile Duct Stone (Hepatobiliary disorders) | 2 | 0
Biliary Colic (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Cholangitis Acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 3 | 3
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 2
Cholelithiasis (Hepatobiliary disorders) | 7 | 5
Cholelithiasis Obstructive (Hepatobiliary disorders) | 0 | 1
Gallbladder Polyp (Hepatobiliary disorders) | 0 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic Lesion (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 1 | 0
Liver Injury (Hepatobiliary disorders) | 0 | 1
Non-Alcoholic Steatohepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic Reaction (Immune system disorders) | 2 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 2 | 1
Abscess Neck (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 2 | 6
Arthritis Bacterial (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 3 | 0
Campylobacter Gastroenteritis (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 11 | 9
Cellulitis Staphylococcal (Infections and infestations) | 0 | 1
Cellulitis Streptococcal (Infections and infestations) | 0 | 1
Cholecystitis Infective (Infections and infestations) | 1 | 1
Colonic Abscess (Infections and infestations) | 0 | 1
Device Related Infection (Infections and infestations) | 1 | 2
Diabetic Foot Infection (Infections and infestations) | 4 | 3
Diabetic Gangrene (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 3 | 3
Ear Infection (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 2
Epididymitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 5 | 0
Escherichia Infection (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 1 | 2
Eye Infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 2 | 5
Gastroenteritis (Infections and infestations) | 9 | 8
Gastroenteritis Viral (Infections and infestations) | 1 | 2
Genital Infection Fungal (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Hiv Infection (Infections and infestations) | 1 | 0
Infected Dermal Cyst (Infections and infestations) | 1 | 0
Infected Skin Ulcer (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 1 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 5
Intervertebral Discitis (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 2
Localised Infection (Infections and infestations) | 6 | 5
Lower Respiratory Tract Infection (Infections and infestations) | 6 | 1
Lung Abscess (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 2 | 0
Osteomyelitis (Infections and infestations) | 5 | 6
Osteomyelitis Chronic (Infections and infestations) | 0 | 1
Otitis Media Acute (Infections and infestations) | 1 | 0
Parasitic Gastroenteritis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 0 | 1
Pelvic Abscess (Infections and infestations) | 1 | 0
Penile Abscess (Infections and infestations) | 0 | 1
Perinephric Abscess (Infections and infestations) | 0 | 1
Peritonsillar Abscess (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 31 | 26
Pneumonia Legionella (Infections and infestations) | 1 | 0
Pneumonia Pneumococcal (Infections and infestations) | 2 | 0
Post Procedural Infection (Infections and infestations) | 0 | 1
Post Procedural Sepsis (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 1
Pulmonary Sepsis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 5
Pyelonephritis Acute (Infections and infestations) | 3 | 1
Respiratory Tract Infection (Infections and infestations) | 13 | 5
Scrotal Abscess (Infections and infestations) | 0 | 1
Scrotal Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 9 | 4
Septic Shock (Infections and infestations) | 6 | 4
Sinusitis (Infections and infestations) | 1 | 0
Soft Tissue Infection (Infections and infestations) | 0 | 2
Staphylococcal Infection (Infections and infestations) | 2 | 0
Staphylococcal Sepsis (Infections and infestations) | 0 | 1
Stenotrophomonas Infection (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 2 | 0
Tooth Abscess (Infections and infestations) | 0 | 1
Tooth Infection (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 2
Urinary Tract Infection (Infections and infestations) | 13 | 11
Urinary Tract Infection Enterococcal (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Wound Infection (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 2 | 0
Arterial Bypass Stenosis (Injury, poisoning and procedural complications) | 0 | 1
Carotid Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 2
Cataract Operation Complication (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 3 | 1
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 2
Epiphyseal Fracture (Injury, poisoning and procedural complications) | 0 | 1
Eye Injury (Injury, poisoning and procedural complications) | 1 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 5
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 6 | 4
Fibula Fracture (Injury, poisoning and procedural complications) | 1 | 2
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 1
Fractured Coccyx (Injury, poisoning and procedural complications) | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 2
Head Injury (Injury, poisoning and procedural complications) | 2 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 5 | 3
Humerus Fracture (Injury, poisoning and procedural complications) | 2 | 3
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0
Limb Crushing Injury (Injury, poisoning and procedural complications) | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 2 | 5
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 1
Meniscus Injury (Injury, poisoning and procedural complications) | 0 | 2
Patella Fracture (Injury, poisoning and procedural complications) | 2 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 1 | 0
Post Laminectomy Syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Haematuria (Injury, poisoning and procedural complications) | 0 | 2
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 2
Postoperative Hernia (Injury, poisoning and procedural complications) | 1 | 0
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 0 | 1
Procedural Headache (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 4 | 4
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 2
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 2
Subarachnoid Haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 | 1
Suture Related Complication (Injury, poisoning and procedural complications) | 0 | 1
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Rupture (Injury, poisoning and procedural complications) | 2 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 1 | 2
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 4
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 2
Traumatic Ulcer (Injury, poisoning and procedural complications) | 1 | 0
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 2
Upper Limb Fracture (Injury, poisoning and procedural complications) | 2 | 1
Vascular Graft Stenosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wound Necrosis (Injury, poisoning and procedural complications) | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriogram Coronary (Investigations) | 2 | 0
Blood Creatinine Increased (Investigations) | 0 | 1
Blood Glucose Increased (Investigations) | 3 | 0
Ejection Fraction Decreased (Investigations) | 1 | 0
Electrocardiogram QT Prolonged (Investigations) | 1 | 0
Electrocardiogram St-T Change (Investigations) | 0 | 1
Electrocardiogram T Wave Inversion (Investigations) | 0 | 1
International Normalised Ratio Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 0 | 1
Platelet Count Decreased (Investigations) | 1 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Diabetes Mellitus (Metabolism and nutrition disorders) | 18 | 5
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 12 | 6
Diabetic Complication (Metabolism and nutrition disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 | 5
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 2 | 1
Gout (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2
Hyperosmolar Hyperglycaemic State (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 2 | 1
Lactic Acidosis (Metabolism and nutrition disorders) | 0 | 2
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 1
Obesity (Metabolism and nutrition disorders) | 3 | 2
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 11 | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Extremity Contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral Disc Compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 5 | 7
Knee Deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 4 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 | 13
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 4
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Spinal Pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 1 | 0
Trigger Finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Adenosquamous Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Benign Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Neoplasm of Thyroid Gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Breast Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral Hygroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 4
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Large Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Lung Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Neoplasm of Unknown Primary Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mediastinum Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to Central Nervous System (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Neuroendocrine Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Papillary Cystadenoma Lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 0
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Serous Cystadenocarcinoma of Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of the Oral Cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ureteric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basilar Artery Occlusion (Nervous system disorders) | 0 | 1
Brain Injury (Nervous system disorders) | 0 | 1
Brain Stem Infarction (Nervous system disorders) | 0 | 1
Brain Stem Stroke (Nervous system disorders) | 0 | 2
Carotid Arteriosclerosis (Nervous system disorders) | 2 | 0
Carotid Artery Occlusion (Nervous system disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 7 | 9
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 1
Cerebellar Infarction (Nervous system disorders) | 1 | 1
Cerebral Haematoma (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 1 | 3
Cerebral Infarction (Nervous system disorders) | 5 | 4
Cerebral Ischaemia (Nervous system disorders) | 1 | 1
Cerebrovascular Accident (Nervous system disorders) | 37 | 15
Cervicobrachial Syndrome (Nervous system disorders) | 1 | 1
Cognitive Disorder (Nervous system disorders) | 1 | 0
Diabetic Mononeuropathy (Nervous system disorders) | 1 | 0
Diabetic Neuropathy (Nervous system disorders) | 1 | 2
Dizziness Postural (Nervous system disorders) | 2 | 2
Embolic Stroke (Nervous system disorders) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 2
Facial Nerve Disorder (Nervous system disorders) | 1 | 0
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 1 | 2
Hemiparesis (Nervous system disorders) | 0 | 2
Hydrocephalus (Nervous system disorders) | 1 | 2
Hypertensive Encephalopathy (Nervous system disorders) | 1 | 0
Hypoxic-Ischaemic Encephalopathy (Nervous system disorders) | 1 | 0
Intraventricular Haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 12 | 20
Lacunar Infarction (Nervous system disorders) | 2 | 2
Lacunar Stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 2
Lumbar Radiculopathy (Nervous system disorders) | 0 | 1
Metabolic Encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Myasthenia Gravis (Nervous system disorders) | 1 | 0
Myasthenia Gravis Crisis (Nervous system disorders) | 0 | 1
Nerve Compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral Nerve Paresis (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 3
Radiculopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 2 | 0
Sensory Loss (Nervous system disorders) | 1 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 8 | 10
Thalamic Infarction (Nervous system disorders) | 0 | 1
Toxic Encephalopathy (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 10 | 8
Tremor (Nervous system disorders) | 0 | 1
Trigeminal Neuralgia (Nervous system disorders) | 0 | 1
Vascular Encephalopathy (Nervous system disorders) | 0 | 1
Vascular Headache (Nervous system disorders) | 1 | 0
Vertebral Artery Occlusion (Nervous system disorders) | 1 | 0
Vertebrobasilar Insufficiency (Nervous system disorders) | 1 | 2
Vocal Cord Paralysis (Nervous system disorders) | 0 | 1
Device Breakage (Product Issues) | 1 | 0
Device Loosening (Product Issues) | 0 | 1
Device Malfunction (Product Issues) | 2 | 0
Patient-Device Incompatibility (Product Issues) | 0 | 1
Bipolar Disorder (Psychiatric disorders) | 2 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Depression Suicidal (Psychiatric disorders) | 0 | 1
Emotional Disorder (Psychiatric disorders) | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 15 | 7
Bladder Obstruction (Renal and urinary disorders) | 0 | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 3
Diabetic Nephropathy (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Ketonuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 8
Nephropathy (Renal and urinary disorders) | 1 | 0
Nephropathy Toxic (Renal and urinary disorders) | 0 | 1
Nephrotic Syndrome (Renal and urinary disorders) | 1 | 0
Pelvi-Ureteric Obstruction (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 2
Renal Failure (Renal and urinary disorders) | 2 | 2
Renal Haematoma (Renal and urinary disorders) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 2 | 1
Renal Injury (Renal and urinary disorders) | 3 | 0
Stress Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 1
Urethral Stenosis (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 2 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 5 | 4
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 1
Endometrial Hypertrophy (Reproductive system and breast disorders) | 1 | 0
Epididymal Disorder (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Fallopian Tube Cyst (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Peyronie's Disease (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 0 | 1
Uterine Prolapse (Reproductive system and breast disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 11 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Vocal Cord Leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 9 | 10
Diabetic Ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Ulcer (Skin and subcutaneous tissue disorders) | 5 | 7
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Penile Prosthesis User (Social circumstances) | 1 | 0
Victim of Homicide (Social circumstances) | 0 | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 1
Hospitalisation (Surgical and medical procedures) | 0 | 1
Stent Placement (Surgical and medical procedures) | 0 | 1
Aortic Aneurysm (Vascular disorders) | 1 | 0
Aortic Arteriosclerosis (Vascular disorders) | 1 | 0
Aortic Stenosis (Vascular disorders) | 4 | 5
Arterial Thrombosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 2
Circulatory Collapse (Vascular disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 2 | 1
Diabetic Vascular Disorder (Vascular disorders) | 1 | 0
Extremity Necrosis (Vascular disorders) | 5 | 3
Haematoma (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 4 | 1
Hypertensive Crisis (Vascular disorders) | 6 | 1
Hypotension (Vascular disorders) | 3 | 0
Hypovolaemic Shock (Vascular disorders) | 0 | 1
Iliac Artery Occlusion (Vascular disorders) | 0 | 1
Intermittent Claudication (Vascular disorders) | 3 | 4
Orthostatic Hypotension (Vascular disorders) | 4 | 1
Peripheral Arterial Occlusive Disease (Vascular disorders) | 9 | 9
Peripheral Artery Occlusion (Vascular disorders) | 1 | 4
Peripheral Artery Stenosis (Vascular disorders) | 2 | 8
Peripheral Artery Thrombosis (Vascular disorders) | 1 | 0
Peripheral Embolism (Vascular disorders) | 1 | 1
Peripheral Ischaemia (Vascular disorders) | 5 | 7
Peripheral Vascular Disorder (Vascular disorders) | 4 | 9
Peripheral Venous Disease (Vascular disorders) | 0 | 1
Poor Peripheral Circulation (Vascular disorders) | 0 | 1
Post Thrombotic Syndrome (Vascular disorders) | 0 | 1
Vascular Insufficiency (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo) (N=2903) | Canagliflozin (Experimental) (N=2904)
Balanoposthitis (Reproductive system and breast disorders) | 25 | 94

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT01989754/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT01989754/SAP_001.pdf